CLINICAL TRIAL: NCT07225699
Title: A SINGLE-CENTER, DOUBLE-ARM, PATIENT MASKED, PROSPECTIVE RANDOMIZED CLINICAL TRIAL TO EVALUATE PATIENT REPORTED OUTCOMES IN PATIENTS WITH CORNEAL ABRASIONS TREATED WITH COLLAGEN CORNEAL SHIELDS IN THE EMERGENCY DEPARTMENT SETTING
Brief Title: IN PATIENTS WITH CORNEAL ABRASIONS TREATED WITH COLLAGEN CORNEAL SHIELDS IN THE EMERGENCY DEPARTMENT SETTING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Murtaza Akhter, Physician Scientist, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00027794
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Corneal Abrasions
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment group (Oasis 72-Hour Collagen Shield) (Experimental): The treatment group will receive an Oasis 72-Hour collagen shield and instructions to take moxifloxacin 0.5% four times daily as well as ibuprofen 400 mg PO q4 hrs as needed for pain.
  Interventions: Device: Oasis 72-Hour collagen shield
- Control Group ( Sham Collagen Shield ) (Active Comparator): The control group will have a sham collagen shield placed (patient will have the impression a lens is placed but it will not actually remain on the eye), and will also be prescribed moxifloxacin 0.5% four times daily and ibuprofen 400 mg PO q4 hrs as needed for pain.
  Interventions: Device: sham collagen shield

INTERVENTIONS:
Device: Oasis 72-Hour collagen shield — All qualified subjects will receive a drop of tetracaine. The treatment group will receive an Oasis 72-Hour collagen shield and instructions to take moxifloxacin 0.5% four times daily as well as ibuprofen 400 mg PO q4 hrs as needed for pain.
  Arms: Treatment group (Oasis 72-Hour Collagen Shield)
Device: sham collagen shield — The control group will have a sham collagen shield placed (patient will have the impression a lens is placed but it will not actually remain on the eye), and will also be prescribed moxifloxacin 0.5% four times daily and ibuprofen 400 mg PO q4 hrs as needed for pain
  Arms: Control Group ( Sham Collagen Shield )

SUMMARY:
This is a single-center, double-arm, patient masked, randomized controlled trial. Subjects will be enrolled in the Emergency Department at the Penn State Milton S. Hershey Medical Center. Eligible subjects must present to the ED and be diagnosed with a traumatic corneal abrasion. One eye from each patient will be considered the study eye.

ELIGIBILITY:
Inclusion Criteria

* Each of the following criteria must be met for study participation:

  1. Male or female, age 18 or older at the time of study enrollment.
  2. Corneal abrasion in one eye.
  3. Willingness to sign the IRB-approved informed consent form (ICF) for study participation.
  4. Availability, willingness, and sufficient cognitive awareness to return for study-required visits and comply with examination procedures.

     Exclusion Criteria:

     Patient candidates presenting any of the following characteristics will not be eligible for study participation:

  <!-- -->

  1. Corneal abrasion in both eyes.
  2. Allergy to moxifloxacin or other fluoroquinolone antibiotics.
  3. Allergy to ibuprofen or other non-steroidal anti-inflammatory drugs.
  4. History of neurotrophic cornea for any reason, in the study eye.
  5. History of medical conditions known to cause decreased corneal sensation in the study eye including but not limited to HSV, HZO, and diabetes.
  6. History of extraocular surgical procedures known to cause decreased corneal sensation in the study eye, including but not limited to trigeminal nerve clamp.
  7. Any anterior segment pathology in the study eye that could significantly affect corneal wound healing (e.g. aniridia, clinically significant corneal dystrophies [ABMD], etc.)
  8. Any visually significant intraocular media opacity other than corneal abrasion in the study eye (as determined by the investigator). Such opacities might include corneal scar or vitreous hemorrhage.
  9. History of any clinically significant retinal pathology or ocular diagnosis in the study eye that could, in the investigator's best judgement, alter or limit visual acuity (e.g. ischemic disease, macular degeneration, retinal detachment, optic neuropathy, amblyopia, strabismus, aniridia, epiretinal membrane, etc.).
  10. History of uveitis in either eye.
  11. History of intraocular or corneal surgery in the study eye besides laser peripheral iridotomy (LPI), retinal barrier laser.
  12. Current ocular infection in the study eye.
  13. Presence of uncontrolled systemic disease that could limit capacity to sign consent or comply with treatment schedule (e.g. mental illness, dementia, etc.).
  14. Unsuitable for study participation for any other reason, as determined by the Investigator's clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score 4 hours | four hours after leaving the emergency department.
  - The primary endpoint will be pain score (10-point Liekert scale) 0=No pain 10=more pain
Pain score 24 hours | 24 hours after discharge from the emergency department
  The Secondary endpoint will be pain score (10-point Liekert scale) score 0=No pain 10=more pain
Pain Score 72 hours | 72 hours after discharge from the emergency department
  The Secondary endpoint will be pain score (10-point Liekert scale) score 0=No pain 10=more pain

SECONDARY OUTCOMES:
Dosage NSAID use in first 24 hours | in the first 24 hours after being discharged from the emergency department
  Dosage of non-steroidal anti-inflammatory drugs (NSAIDs)
Frequency NSAID 24 Hour | 24 Hour
Pain score 24 hours | 24 hours after discharge from the emergency department
  The Secondary endpoint will be pain score (10-point Liekert scale) score 0=No pain 10=more pain

CONTACTS AND LOCATIONS:
Overall Officials: Murtaza Akhter, MD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No